CLINICAL TRIAL: NCT05942846
Title: POLECAT: Perioperative Delta Renin Concentration
Acronym: POLECAT
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Royal Surrey County Hospital NHS Foundation Trust (Other)
Collaborators: European Society of Intensive Care Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: 319836
Record Dates: First submitted 2023-07-04; First posted 2023-07-12 (Actual); Last update posted 2023-07-12 (Actual); Status verified 2023-07

CONDITIONS: Post Operative Vasoplegic Syndrome; Acute Kidney Injury
MeSH Terms: conditions — Vasoplegia; Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — • Ethylenediaminetetraacetic acid (EDTA) blood bottles will be centrifuged using a refrigerated centrifuge for 15 minutes to separate the plasma.
  . PAXGene for subsequent leukocyte transcriptomics analysis.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
We want to measure the amount of a hormone called renin in people's bodies before and after they have major abdominal surgery. We want to see if changes in renin levels are connected to problems with blood flow, unstable blood pressure, and kidney damage after surgery.

DETAILED DESCRIPTION:
The renin-angiotensin system (RAS) plays a key role in haemodynamic stability, vascular tone and electrolyte homeostasis. It is recognised that this system is dysfunctional during critical illness. It remains unknown as to whether significant dysfunction of RAS is found in patients who have undergone major abdominal surgery - however over 50% of these patients often require blood pressure support post-operatively, with nearly half of these patients having unexplained drops in blood pressure.

Renin represents an attractive biomarker that could be implicated in post operative vasoplegia and post operative AKI and as such elevated renin concentrations could be used to identify high-risk patients for cardiovascular instability and AKI who would benefit from timely intervention that could improve their outcomes, this would include the use of selective vasopressor agents such as angiotensin II which has been shown to confer a benefit in patients with underlying dysregulation of the RAS.

If we show that higher differences in renin concentrations are associated with a greater incidence of vasoplegia then we can design a subsequent clinical trial with a different treatment in those who have a higher change in renin. Such a trial is currently recruiting in Germany for patients with higher changes in renin due to cardiac surgery.

The primary aim is to assess whether there is an association between higher differences in renin concentrations (a protein that can be measured in your blood) and haemodynamic instability manifest as vasoplegia (patients exhibiting low blood pressure) in patients undergoing major abdominal surgery requiring post-operative admission to ICU.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* All patients having abdominopelvic surgery (planned or unplanned) needing ICU admission where arterial line or central line will been placed
* Able to provide consent, or personal/professional agreement

Exclusion Criteria:

* Patient < 18 years old at time of screening
* Patients already receiving vasopressor support pre-operatively
* Receiving palliative care at the time of recruitment or expected to die within next 24 hours
* Those on kidney replacement therapy (KRT) or end stage kidney disease (ESKD)
* Patient or consultee unable to communicate in verbal and written English
* Patients held in an institution by legal or official order
* Patients with severe mental health disorders that might impair their capacity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Planned and unplanned emergency general surgical procedures. All surgical patients who have an intensive care bed booked, will be screened.
  To sample patients we will approach all patients who are booked to come to the ICU post operatively.
Sampling Method: Non-Probability Sample
Enrollment: 405 (Estimated)
Dates: Start 2023-07 (Estimated); Primary Completion 2025-07 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
• The difference between pre and post-operative levels of circulating renin, and association with vasoplegia. | 2 years

SECONDARY OUTCOMES:
• Determine overall burden of vasopressor use post operatively. | 2 years
• Incidence of post-operative AKI in this cohort of patients | 2 years
• Trends of renin post-operatively following major abdominal surgery. | 2 years
• Associations between changes in renin and AKI. | 2 years
• Associations between type of surgery and incidence of post operative instability and renin measurements, with specific emphasis on patients with emergency surgery with peritonitis. | 2 years
• Association between regular medications that alter the RAS-axis and changes in renin | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Lui Forni, Principal Investigator — Professor of Intensive Care Medicine, Royal Surrey Hospital